CLINICAL TRIAL: NCT07119021
Title: Efficacy and Safety Study of Ultra-early Mobile Stroke Unit Neuroprotection Combined With Revascularization for Acute Ischemic Stroke (EXCELLENT)
Acronym: EXCELLENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijun Ji (Other)
Collaborators: Xing'an League People's Hospital (Unknown); Suzhou First People's Hospital (Unknown); Nanyang nanshi Hospital (Unknown); Nanjing Baixinyu Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Ruijun Ji, Chief Physician/Professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023ZD0503805; NS&T(2023ZD0503805) (Other: Medicine and Health Science and Technology Development Research Center of the National Health Commission)
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: Acute Ischemic Stroke; Bleeding Conversion; Edaravone Sublingual Tablets
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone; Fibrinolytic Agents; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous thrombolysis + edaravone (intervention group) (Experimental): The patient underwent intravenous t-PA thrombolysis and sublingual administration of edaravone tablets in the prehospital ambulance. The method of intravenous t-PA thrombolysis is in accordance with the international guidelines: t-PA dose is calculated according to 0.9mg/kg; 10% of the total dose is injected intravenously, and the remaining 90% is administered intravenously at a uniform rate within one hour.
  Interventions: Drug: Intravenous thrombolysis + edaravone
- IV thrombolysis + placebo (control group) (Placebo Comparator): Patients underwent intravenous t-PA thrombolysis + placebo sublingual administration. The method of intravenous t-PA thrombolysis is in accordance with the international guideline standards: t-PA dose is calculated according to 0.9mg/kg; 10% of the total dose is injected intravenously, and the remaining 90% is administered intravenously at a constant rate within 1 hour.
  Interventions: Drug: IV thrombolysis + placebo (control group)

INTERVENTIONS:
Drug: Intravenous thrombolysis + edaravone — The patient underwent intravenous t-PA thrombolysis and sublingual administration of edaravone tablets in the prehospital ambulance. Intravenous t-PA thrombolysis was performed in accordance with international guidelines: t-PA dose was calculated according to 0.9mg/kg; 10% of the total dose was injected intravenously, and the remaining 90% was administered intravenously at a uniform rate within one hour.
  Arms: Intravenous thrombolysis + edaravone (intervention group)
Drug: IV thrombolysis + placebo (control group) — Patients underwent intravenous t-PA thrombolysis + placebo sublingual administration. The method of intravenous t-PA thrombolysis is in accordance with the international guideline standards: t-PA dose is calculated according to 0.9mg/kg; 10% of the total dose is injected intravenously, and the remaining 90% is administered intravenously at a constant rate within 1 hour.
  Arms: IV thrombolysis + placebo (control group)

SUMMARY:
EXCELLENT was a prospective, multicenter, randomized, double-blind, placebo-controlled clinical study in which participants were randomized participants were randomized (1:1) to receive either IV thrombolysis + edaravone or IV thrombolysis + matched placebo (same volume of tablets without drug components), and the primary outcome was the proportion of patients with transformed bleeding on MRI at 72 hours following revascularization therapy.

DETAILED DESCRIPTION:
1. Study on the effectiveness of neuroprotection combined with revascularization in the treatment of acute ischemic stroke in the ultra-early mobile stroke unit (MSU):

   Based on the MSU model, using the RCT study design, for patients with disabling AIS within 4.5h, patients were randomly assigned 1:1 to the experimental group and the control group and were given the neuroprotective agent edaravone tablets + intravenous thrombolysis and placebo + intravenous thrombolysis interventions, respectively. The main evaluation index was the proportion of patients with transformed blood flow on MRI at 72 hours after receiving recanalization, and the other indexes included the patients' 90-day onset The remaining indicators include the modified Rankin Scale (mRS) score (hierarchical data), the proportion of patients with an mRS score of <1 at 90 days of onset, the proportion of patients with an mRS score of <2 at 90 days of onset, the time from onset to intravenous thrombolysis (in minutes), and the proportion of patients who received intravenous thrombolysis within 60 minutes of onset.
2. Safety study of ultra-early mobile stroke unit neuroprotection combined with revascularization for acute ischemic stroke:

Based on the MSU model, using the RCT study design for patients with disabling AIS within 4.5h, patients were 1:1 randomly assigned to the experimental group and control group, and were given the neuroprotective agent edaravone tablets + intravenous thrombolysis and placebo + intravenous thrombolysis interventions, respectively. The main safety evaluation indexes included all deaths during hospitalization, hospitalized deaths after receiving intravenous thrombolysis, deaths at 3 months after stroke, deaths at 3 months after receiving intravenous thrombolysis, and the proportion of symptomatic intracranial hemorrhage within 36 hours of the onset of the disease, and so on.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Acute ischemic stroke as defined by the International Health Organization (WHO) and confirmed by cranial CT;
* Onset within a 4.5-hour time window;
* NIHSS score of 6-24;
* Meet the criteria for intravenous thrombolysis in acute ischemic stroke recommended by international guidelines;
* Patient or family consent.

Exclusion Criteria:

* Pregnant women, women in labor, and patients in the puerperium;
* Comorbidity with other serious diseases that affect outcome determination;
* Comorbidity with other serious diseases that affect prognostic regression;
* Comorbidity with other serious diseases with a life expectancy of less than 1 year;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint indicators | From the start of revascularization until 72 hours after treatment.
  Proportion of patients with transformed bleeding on MRI at 72 hours after revascularization.

SECONDARY OUTCOMES:
Secondary endpoint indicators | 90 days after onset of illness
  1. Patients' modified Rankin Scale (mRS) scores at 90 days after onset of illness (hierarchical data).
     (i) Proportion of patients with mRS score <1 at 90 days of disease onset; (ii) Proportion of patients with mRS score <2 at 90 days of presentation;
  2. Time from onset to intravenous thrombolytic therapy (in minutes);
  3. Proportion of patients receiving intravenous thrombolytic therapy within 60 minutes of onset;
  4. Proportion of patients receiving subsequent endovascular treatment;
  5. Time from onset to femoral artery puncture (minutes);

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No